CLINICAL TRIAL: NCT04088656
Title: Systems Analysis and Improvement Approach to Optimize the Hypertension Diagnosis and Care Cascade for HIV-infected Individuals
Brief Title: Systems Analysis and Improvement Approach for the Hypertension Care Cascade
Acronym: SAIA-HTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sarah Odell Gimbel-Sherr, Associate Professor, School of Nursing: Family and Child Nursing, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006694; R01HL142412 (NIH)
Record Dates: First submitted 2019-07-01; First posted 2019-09-13 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: HIV/AIDS; Hypertension
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertension Systems Analysis and Improvement (Experimental): Eight (8) health facilities will receive the Systems Analysis and Improvement Approach (SAIA-HTN) intervention to optimize hypertension screening and management for people living with HIV/AIDS.
  Interventions: Other: Systems Analysis and Improvement Approach for Hypertension Screening and Treatment Optimization
- Control (No Intervention): Eight (8) health facilities will not receive the Systems Analysis and Improvement Approach (SAIA-HTN) intervention to optimize hypertension screening and management for people living with HIV/AIDS.

INTERVENTIONS:
Other: Systems Analysis and Improvement Approach for Hypertension Screening and Treatment Optimization — The Systems Analysis and Improvement Approach to Optimize the Hypertension Care Cascade for People Living with HIV (SAIA-HTN) is a five-step systems analysis and iterative improvement cycle intervention which will be implemented by study nurses and district managers in intervention facilities. Components of the intervention include joint care cascade analysis, patient flow mapping and continuous quality improvement, aimed to incrementally improve hypertension screening, diagnosis, treatment and care in the HIV+ population at intervention health facilities.
  Arms: Hypertension Systems Analysis and Improvement

SUMMARY:
As undiagnosed and untreated hypertension is one of the largest drivers of cardiovascular disease in sub-Saharan Africa approaches are needed to optimize the hypertension care cascade. The HIV treatment platform in low and middle income countries provides a robust, scalable foundation to address other chronic care priorities, such as hypertension. This proposal will evaluate an evidence-based intervention designed to improve chronic care services (the Systems Analysis and Improvement Approach (SAIA)) for hypertension detection and management in people living with HIV, and will build evidence on how to achieve rapid, sustainable and scalable improvements in services that can dramatically improve population health in resource-limited countries.

ELIGIBILITY:
Inclusion Criteria:

* (A1) Frontline Health Workers / Health Facility Managers currently working in outpatient, emergency or related (pharmacy, laboratory) services at one of the study clinics in Manica and Sofala provinces, Mozambique; (A2) District Health Supervisors currently employed in a study district in Manica and Sofala provinces, Mozambique regularly engaged in service provision or management of HIV-infected and/or hypertensive populations; and (A3) Clinical Experts currently working in Mozambique in the clinical delivery of HIV and/or hypertension care and treatment or (B1) People Living with HIV >14 years old (B2) access HIV care and treatment services via outpatient/emergency services in study clinics. >14 years is being used as the current Ministry of Health forms only use the age bounds of <15y, >14y and there is significant concern by the Mozambican Ministry of Health to minimize additional data collection when not absolutely necessary.

Exclusion Criteria:

* (A1) not currently working as a Frontline Health Worker/Health Facility Manager at a participating study facility or (A2) not currently working as a District Health Supervisor in a participating district or (A3) not currently working in Mozambique in the clinical delivery of HIV and/or hypertension care and treatment or (B1) HIV-negative or of unknown status or (B2) <15 years old or age not recorded, (B3) or pregnant or postpartum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah O Gimbel-Sherr, RN, PhD, MPH, Principal Investigator — University of Washington
Locations (16):
- Mozambique (16):
  - Hospital Distrital de Catandica, Catandica, Manica Province
  - Centro de Saude 1 de Maio, Chimoio, Manica Province
  - Centro de Saude 7 de Abril, Chimoio, Manica Province
  - Centro de Saude Eduardo Mondlane, Chimoio, Manica Province
  - Centro de Saude Nhamaonha, Chimoio, Manica Province
  - Centro de Saude de Sussundenga, Sussundenga, Manica Province
  - Centro de Saude Vanduzi, Vanduzi, Manica Province
  - Centro de Saude de Macurungo, Beira, Sofala
  - Centro de Saude de Manga Mascarenhas, Beira, Sofala
  - Centro de Saude de Manga Nhanconjo, Beira, Sofala
  - Centro de Saude de Ponte Gea, Beira, Sofala
  - Hospital Rural de Buzi, Búzi, Sofala
  - Centro de Saude de Dondo, Dondo, Sofala
  - Centro de Saude de Mafambisse, Dondo, Sofala
  - Hospital Rural de Nhamatanda, Nhamatanda, Sofala
  - Hospital Distrital de Manica, Manica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gimbel S, Mocumbi AO, Asbjornsdottir K, Coutinho J, Andela L, Cebola B, Craine H, Crocker J, Hicks L, Holte S, Hossieke R, Itai E, Levin C, Manaca N, Murgorgo F, Nhumba M, Pfeiffer J, Ramiro I, Ronen K, Sotoodehnia N, Uetela O, Wagner A, Weiner BJ, Sherr K. Systems analysis and improvement approach to optimize the hypertension diagnosis and care cascade for PLHIV individuals (SAIA-HTN): a hybrid type III cluster randomized trial. Implement Sci. 2020 Mar 6;15(1):15. doi: 10.1186/s13012-020-0973-4. PMID 32143657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We randomly allocated health facilities (n=16) to the intervention (n=8) or control (n=8). We consented healthcare workers for qualitative interviews and surveys (n=305) throughout the study. There is no interaction with patients (patients are not consented nor enrolled), however we use the clinical outcomes of patients to determine the effect our implementation strategy (SAIA-HTN). Patient-level data comes from routine data sources and is de-identified. Data from 65,625 patients were captured.
Units Other Than Participants: health facilities
Period: Baseline Period
Arm/Group | Hypertension Systems Analysis and Improvement | Control
Started | 12307; 8 health facilities | 10042; 8 health facilities
Patients | 12307; 8 health facilities | 10042; 8 health facilities
Completed | 12307; 8 health facilities | 10042; 8 health facilities
Not Completed | 0; 0 health facilities | 0; 0 health facilities
Period: Intensive Implementation Period
Arm/Group | Hypertension Systems Analysis and Improvement | Control
Started | 20788; 8 health facilities (Patients were counted in the phase in which they first came to the facility to receive HIV care. If they were captured in the previous period, they were not counted in this period or the subsequent period.) | 17909; 8 health facilities (Patients were counted in the phase in which they first came to the facility to receive HIV care. If they were captured in the previous period, they were not counted in this period or the subsequent period.)
Healthcare Workers | 171; 8 health facilities | 0; 0 health facilities (In the control sites, the SAIA-HTN intervention was not delivered and thus there were no healthcare workers enrolled as they didn't receive the intervention.)
Patients (Patients were counted in the phase in which they first came to the facility to receive HIV care. If they were captured in the previous period, they were not counted in this period or the subsequent period.) | 20617; 8 health facilities | 17909; 8 health facilities
Completed | 20788; 8 health facilities | 17909; 8 health facilities
Not Completed | 0; 0 health facilities | 0; 0 health facilities
Period: Sustainment Implementation Period
Arm/Group | Hypertension Systems Analysis and Improvement | Control
Started | 2317; 8 health facilities (Patients were counted in the phase in which they first came to the facility to receive HIV care. If they were captured in the previous period, they were not counted in this period.) | 2567; 8 health facilities (Patients were counted in the phase in which they first came to the facility to receive HIV care. If they were captured in the previous period, they were not counted in this period.)
Healthcare Workers | 134; 8 health facilities | 0; 0 health facilities (In the control sites, the SAIA-HTN intervention was not delivered and thus there were no healthcare workers enrolled as they didn't receive the intervention.)
Patients (Patients were counted in the phase in which they first came to the facility to receive HIV care. If they were captured in the previous period, they were not counted in this period.) | 2183; 8 health facilities | 2567; 8 health facilities
Completed | 2317; 8 health facilities | 2567; 8 health facilities
Not Completed | 0; 0 health facilities | 0; 0 health facilities

BASELINE CHARACTERISTICS:
Population: Enrolled and consented 305 healthcare workers in intervention sites and none in control sites. Data captured from 35107 patients in intervention sites and 30518 control sites.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypertension Systems Analysis and Improvement | Control | Total
Number analyzed (Participants) | 35412 | 30518 | 65930
Age, Categorical [Count of Participants; unit: Participants] — Population: We consent healthcare workers for qualitative collection (n=305) throughout the study. There is no interaction with patients (patients are not consented nor enrolled), however we use the clinical outcomes of patients to determine the effect of SAIA-HTN. Patient-level data comes from routine data sources and is de-identified. Data from 65,625 patients were captured. Age is missing for 52 patients in control sites and 966 patients in intervention sites.
  Participants
    Healthcare Workers: number analyzed (Participants) | 305 | 0 | 305
    Healthcare Workers: <=18 years | 0 | 0 | 0
    Healthcare Workers: Between 18 and 65 years | 305 | 0 | 305
    Healthcare Workers: >=65 years | 0 | 0 | 0
    Patients: number analyzed (Participants) | 34141 | 30466 | 64607
    Patients: <=18 years | 0 | 0 | 0
    Patients: Between 18 and 65 years | 33465 | 29871 | 63336
    Patients: >=65 years | 676 | 595 | 1271
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We consent healthcare workers for qualitative collection (n=305) throughout the study. Sex is missing for 21 healthcare workers. There is no interaction with patients (patients are not consented nor enrolled), however we use the clinical outcomes of patients to determine the effect of SAIA-HTN. Patient-level data comes from routine data sources and is de-identified. Data from 65,625 patients were captured. Sex is missing for 10 patients in control sites and 28 patients in intervention sites.
  Participants
    Healthcare Workers: number analyzed (Participants) | 284 | 0 | 284
    Healthcare Workers: Female | 132 | 0 | 132
    Healthcare Workers: Male | 152 | 0 | 152
    Patients: number analyzed (Participants) | 35079 | 30508 | 65587
    Patients: Female | 22718 | 18821 | 41539
    Patients: Male | 12361 | 11687 | 24048
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We consent healthcare workers for qualitative collection (n=305) throughout the study. There is no interaction with patients (patients are not consented nor enrolled), however we use the clinical outcomes of patients to determine the effect of SAIA-HTN. Patient-level data comes from routine data sources and is de-identified. Data from 65,625 patients were captured.
  Participants
    Healthcare Workers: number analyzed (Participants) | 305 | 0 | 305
    Healthcare Workers: American Indian or Alaska Native | 0 | 0 | 0
    Healthcare Workers: Asian | 0 | 0 | 0
    Healthcare Workers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Healthcare Workers: Black or African American | 305 | 0 | 305
    Healthcare Workers: White | 0 | 0 | 0
    Healthcare Workers: More than one race | 0 | 0 | 0
    Healthcare Workers: Unknown or Not Reported | 0 | 0 | 0
    Patients: number analyzed (Participants) | 35107 | 30518 | 65625
    Patients: American Indian or Alaska Native | 0 | 0 | 0
    Patients: Asian | 0 | 0 | 0
    Patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Patients: Black or African American | 35107 | 30518 | 65625
    Patients: White | 0 | 0 | 0
    Patients: More than one race | 0 | 0 | 0
    Patients: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Healthcare workers and Patients]
  Mozambique | 35412 | 30518 | 65930

OUTCOME MEASURES:

1. Primary Outcome: Controlled Hypertension
Description: The proportion of HIV-infected patients with controlled hypertension among those who were diagnosed with hypertension and picked up their medications after receiving a prescription
Time Frame: Per Phase: up 3 months for Baseline Phase, up to 2 years for Intensive Implementation Phase, up to 1 year for Sustainment Phase.
Population: Number of new and existing HIV-infected patients attending enrolled facilities who were diagnosed with hypertension and picked up their medications after receiving a prescription
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Arm - Baseline Phase: Newly eligible HIV-infected patients attending intervention facilities during baseline phase
- Intervention Arm - Intensive Implementation Phase: Newly eligible HIV-infected patients attending intervention facilities during intensive implementation phase
- Intervention Arm - Sustainment Phase: Newly eligible HIV-infected patients attending intervention facilities during sustainment phase
- Control Arm - Baseline Phase: Newly eligible HIV-infected patients attending control facilities during baseline phase
- Control Arm - Intensive Implementation Phase: Newly eligible HIV-infected patients attending control facilities during intensive implementation phase
- Control Arm - Sustainment Phase: Newly eligible HIV-infected patients attending control facilities during sustainment phase
Arm/Group | Intervention Arm - Baseline Phase | Intervention Arm - Intensive Implementation Phase | Intervention Arm - Sustainment Phase | Control Arm - Baseline Phase | Control Arm - Intensive Implementation Phase | Control Arm - Sustainment Phase
Number analyzed (Participants) | 74 | 1447 | 157 | 52 | 1430 | 161
Participants | 3 | 315 | 37 | 1 | 82 | 14

2. Secondary Outcome: Blood Pressure Screening
Description: The proportion of HIV-infected patients who were screened for hypertension
Time Frame: as for outcome 1
Population: Number of new and existing HIV-infected patients attending enrolled facilities
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm - Baseline Phase | Intervention Arm - Intensive Implementation Phase | Intervention Arm - Sustainment Phase | Control Arm - Baseline Phase | Control Arm - Intensive Implementation Phase | Control Arm - Sustainment Phase
Number analyzed (Participants) | 12307 | 20617 | 2183 | 10042 | 17909 | 2567
Participants | 4275 | 20359 | 2182 | 3351 | 17882 | 2556

3. Secondary Outcome: Hypertension Diagnosis
Description: The proportion of HIV-infected patients diagnosed with hypertension among those who were screened
Time Frame: as for outcome 1
Population: Number of new and existing HIV-infected patients attending enrolled facilities who were screened for hypertension
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm - Baseline Phase | Intervention Arm - Intensive Implementation Phase | Intervention Arm - Sustainment Phase | Control Arm - Baseline Phase | Control Arm - Intensive Implementation Phase | Control Arm - Sustainment Phase
Number analyzed (Participants) | 4275 | 20359 | 2182 | 3351 | 17882 | 2556
Participants | 318 | 2247 | 244 | 288 | 2442 | 404

4. Secondary Outcome: Hypertension Treatment Prescription
Description: The proportion of hypertension medication-eligible HIV patients receiving a prescription
Time Frame: as for outcome 1
Population: Number of new and existing HIV-infected patients attending enrolled facilities who were diagnosed with hypertension (i.e. medication-eligible)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm - Baseline Phase | Intervention Arm - Intensive Implementation Phase | Intervention Arm - Sustainment Phase | Control Arm - Baseline Phase | Control Arm - Intensive Implementation Phase | Control Arm - Sustainment Phase
Number analyzed (Participants) | 318 | 2247 | 244 | 288 | 2442 | 404
Participants | 221 | 1678 | 177 | 175 | 1698 | 256

5. Secondary Outcome: Hypertension Medication Pick up
Description: The proportion of HIV patients who are hypertension medication-eligible and pick up their medications after receiving a prescription
Time Frame: as for outcome 1
Population: Number of new and existing HIV-infected patients attending enrolled facilities who were diagnosed with hypertension (i.e. medication-eligible) and prescribed hypertension medication
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm - Baseline Phase | Intervention Arm - Intensive Implementation Phase | Intervention Arm - Sustainment Phase | Control Arm - Baseline Phase | Control Arm - Intensive Implementation Phase | Control Arm - Sustainment Phase
Number analyzed (Participants) | 221 | 1678 | 177 | 175 | 1698 | 256
Participants | 74 | 1447 | 157 | 52 | 1430 | 161

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years.
Description: Definition of adverse event / serious adverse event does not differ from that of clinicaltrials.gov. Adverse Events were only monitored/assessed in healthcare worker participants. No healthcare worker participants were at risk in the control arm as no intervention was applied and thus no healthcare workers were exposed or at risk. All-Cause Mortality, Serious Adverse Events, and Other Adverse Events were not monitored/assessed in patient participants.
Arm/Group | Hypertension Systems Analysis and Improvement | Control
All-Cause Mortality (participants affected / at risk) | 0/305 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/305 | 0/0
Other Adverse Events (participants affected / at risk) | 0/305 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04088656/Prot_SAP_000.pdf